CLINICAL TRIAL: NCT06212128
Title: Novel Objective Comparison of Short-term Surgical Outcomes From Total Mesorectal Excision Between Total Neoadjuvant Therapy - Rapido Protocol, Standard Long Course Radiotherapy and Upfront Surgery
Brief Title: RAPIDO vs LCRT vs Upfront Surgery - a Prospective Cohort Study
Acronym: RAPIDO
Status: Active, not recruiting | Type: Observational
Sponsor: Sengkang General Hospital (Other)
Responsible Party: Principal Investigator, Koh Hong Xiang Frederick, Consultant, Sengkang General Hospital
Other Study IDs: CIRB: 2020/2525
Record Dates: First submitted 2023-12-27; First posted 2024-01-18 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Surgical outcomes; Neoadjuvant treatment
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RAPIDO TNT: neoadjuvant therapy per RAPIDO protocol
  Interventions: Combination Product: RAPIDO TNT
- LCRT: long course chemoradiotherapy
  Interventions: Combination Product: LCRT
- upfront surgery: directly went for surgery after diagnosis of rectal cancer

INTERVENTIONS:
Combination Product: RAPIDO TNT — neoadjuvant therapy per RAPIDO protocol (Patients under RAPIDO group underwent 25Gy/5 sessions of short course radiotherapy followed by 6 cycles of neoadjuvant XELOX similar to that of the RAPIDO trial protocol)
  Groups: RAPIDO TNT
Combination Product: LCRT — LCRT group underwent conventional 50Gy/25-28 sessions of long course radiotherapy with concurrent oral capecitabine
  Groups: LCRT

SUMMARY:
Aim: We evaluated the surgical outcomes of 3 groups of patients with rectal cancers - RAPIDO vs standard long course radiotherapy (LCRT) vs upfront surgery to objectively determine the effects of TNT on TME.

Methods: A review of prospectively collected data was performed for patients who have rectal cancer and underwent low anterior resection from January 2016 to May 2022. Data on patient demographics, disease staging, peri-operative details and up to 2-year follow-up outcomes were analysed. The surgical and oncological outcomes were compared. Patients were followed up until 31 May 2022.

DETAILED DESCRIPTION:
A review of prospectively collected data was performed for all patients who were diagnosed with rectal cancer and who underwent ultra-low anterior resection (ULAR) from January 2016 to May 2022 in a single institution in Singapore. Exclusion criteria of this study included patients who underwent emergency surgery and patients with unresectable metastatic disease at presentation. All patients were discussed at multi-disciplinary tumour board for recommendation and decision of the respective treatment protocols. Patients were analysed in 3 main categories: neoadjuvant therapy per RAPIDO protocol, LCRT and upfront surgery. Patients under RAPIDO group underwent 25Gy/5 sessions of short course radiotherapy followed by 6 cycles of neoadjuvant XELOX similar to that of the RAPIDO trial protocol while patients in LCRT group underwent conventional 50Gy/25-28 sessions of long course radiotherapy with concurrent oral capecitabine. All cases were performed by 7 consultant-grade colorectal surgeons in the department.

Patient demographics and peri-operative details were collected. Histopathological stage of disease was in accordance with the American Joint Committee on Cancer (AJCC) staging manual after surgical resection with review of the resected specimen by consultant-grade pathologists who were blinded to the type of pre-operative treatment the patients received.

Primary outcome for the study was the operative time required for primary resection of rectal tumour. If combined surgery was performed for oligometastatic disease, we removed the operating time for non-rectal component as this was separately defined in the operation notes.

Secondary outcomes included the intraoperative blood loss, duration to stoma function, failure to remove urinary catheter, presence of post-operative ileus, duration of hospitalisation after surgery. Presence of stoma function was defined as enteric content of significant amount (>200ml or presence of formed faecal material). Failure of removal of urinary catheter is defined as acute urinary retention requiring re-insertion of catheter post-operatively. Post-operative ileus is defined as ileus which persist beyond 7 days from operation.

Follow-up outcomes and data for patients were collected until 31 May 2022. Local-regional recurrence was defined as the first clinical, radiologic and/or pathologic evident tumour of the same histological type at the region of the anastomosis and pelvis. Distant recurrent was defined similarly at sites outside primary malignancy such as liver, lung, bone, brain, para-aortic region. Presence of recurrence in patients was recorded, disease-free interval was calculated in months from date of surgery to date of recurrence.

Statistical analysis All data was analysed with SPSS version 28 (SPSS Inc, Chicago, III). Patients with missing data were accounted for and excluded during the statistical analysis of this data. Categorical variables were presented as percentages while median and interquartile ranges were presented for continuous variables. Differences between categorical variables were analysed using either Chi-square or Student t-test. Differences between continuous variables were treated as non-parametric and analysed using either Kruskal Willis or Mann-Whitney U. Two-sided tests were used, with p value <0.05 treated as significant. Kaplan Meier curves were plotted for survival data including disease free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with rectal cancer
* due to undergo ultra-low anterior resection (ULAR)

Exclusion Criteria:

* emergency surgery
* unresectable metastatic disease at presentation

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: as above
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
operative time required for primary resection of rectal tumour | 1 day
  operative time in minutes

SECONDARY OUTCOMES:
intraoperative blood loss | 30 days post surgery
  in ml
duration to stoma functioning | 14 days post surgery
  in days
failure to remove urinary catheter | 14 days post surgery
  yes/no, and in days to successful removal
presence of post op ileus (defined as >7 days intolerance to diet or no stoma output from time of operation) | 14 days post surgery
  yes/no
duration of hospitalisation | 30 days after surgery
  in days from time of surgery

IPD SHARING:
Plan to Share IPD: Undecided